CLINICAL TRIAL: NCT05195814
Title: An Investigation of Tofacitinib PsA Initiators in the CorEvitas SpA Registry
Brief Title: A Study to Learn About the Study Medicine (Called Tofacitinib) in People With Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3921411
Record Dates: First submitted 2021-12-21; First posted 2022-01-19 (Actual); Results first posted 2025-03-30 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Effectiveness of tofacitinib: Participants receiving tofacitinib will be included to assess the effectiveness of tofacitinib overall and stratified by key variables of interest

SUMMARY:
The purpose of this study is to learn about the safety and effects of the study medicine for the potential treatment of Psoriatic Arthritis (PsA). Psoriatic Arthritis is a joint swelling disease that can also affect the skin, nails and eyes. The study medicine is called Tofacitinib. This study is seeking participants who:

* Started taking tofacitinib alone or with other approved medicines (eg. methotrexate, leflunomide, sulfasalazine, apremilast) for PsA disease. We will only look at participants' who started tofacitinib after December 14, 2017.
* Have a 6-month follow-up visit (with a 3-month window) This is an observational study. Participants receiving Tofacitinib will be included to assess how well tofacitinib works. We will look at participants' demographic information and therapy history. We will also monitor participants' disease progression before and 6 months after treatment. We will examine the experiences of people receiving the study medicine. This will help us determine if the study medicine is safe and effective.

DETAILED DESCRIPTION:
Tofacitinib is an oral Janus kinase (JAK) inhibitor approved in 2017 by the US Food and Drug Administration (FDA) for the treatment of adult patients with active PsA who have had an inadequate response or intolerance to methotrexate or other disease modifying antirheumatic drugs (DMARDs). As of December 3, 2021, Tofacitinib is approved for use in patients who have had an inadequate response or intolerance to one or more TNF blockers.

This is an observational retrospective cohort study that will be conducted using patients enrolled in the CorEvitas PsA/SpA Registry, initiating tofacitinib on or after December 14th, 2017. Patients receiving tofacitinib will be included to assess the effectiveness of tofacitinib overall and when stratified by key variables of interest. More specifically, the overall aim will be to describe baseline demographic, therapy history, and disease activity characteristics and assess change in disease activity measures six months after initiation of tofacitinib.

There are two primary objectives for this study:

1. To describe the effectiveness of all tofacitinib initiators at 6 months in PsA patients
2. To describe the effectiveness of all tofacitinib initiators at 6 months stratified by monotherapy and combination therapy of PsA

ELIGIBILITY:
Inclusion Criteria:

* PsA patients in CorEvitas initiating tofacitinib monotherapy or in combination with oral small molecules (eg methotrexate, leflunomide, sulfasalazine, apremilast) after 14 December 2017 (market approval of tofacitinib in the US) with no prior use of tofacitinib. Only the patient's first initiation after December 14, 2017 will be included in the analysis
* Have a 6 month follow-up visit (with ±3 month window)

Exclusion Criteria:

* Patients taking tofacitinib in combination with any other bDMARD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in an existing registry database
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Ogdie A, Middaugh N, Blachley T, Bourgeois T, Ling YL, Mundayat R, Fallon L, Masri KR, Mease PJ. Effectiveness of Tofacitinib in Patients with Psoriatic Arthritis Initiating Monotherapy Versus Combination Therapy: Results from the CorEvitas Psoriatic Arthritis/Spondyloarthritis Registry. Rheumatol Ther. 2026 Feb;13(1):195-212. doi: 10.1007/s40744-025-00811-4. Epub 2025 Dec 4. PMID 41343116
- [Derived] Mease PJ, Young P, Fallon L, Mundayat R, Dina O, Blachley T, Middaugh N, Ogdie A. Effectiveness of Tofacitinib in Patients Initiating Therapy for Psoriatic Arthritis: Results from the CorEvitas Psoriatic Arthritis/Spondyloarthritis Registry. Rheumatol Ther. 2024 Apr;11(2):313-329. doi: 10.1007/s40744-023-00631-4. Epub 2024 Jan 22. PMID 38252211
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921411

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study included data from CorEvitas Psoriatic Arthritis/ Spondyloarthritis (PsA/SpA) registry.
Pre-assignment Details: A total of 141 PsA participants who initiated tofacitinib monotherapy or in combination with oral small molecules (OSM) (example: methotrexate, leflunomide, sulfasalazine, apremilast) on or after 14-Dec-2017 to 31-August-2023, with no prior use of tofacitinib were included in this study. Data was evaluated over 23.5 months in this retrospective observational study.
Groups:
- Tofacitinib Monotherapy: All participants with a diagnosis of PsA/SpA who received tofacitinib monotherapy with no other (pre-existing or new) disease modifying antirheumatic drug (DMARD) prescriptions on or after 14 December 2017 and had a 6-month follow-up visit were included in this retrospective observational study.
- Tofacitinib + OSM Combination Therapy: All participants with a diagnosis of PsA/SpA who received tofacitinib with a concomitant (pre-existing or new) prescription of at least one OSM (methotrexate, leflunomide, sulfasalazine, apremilast) on or after 14 December 2017 and had a 6-month follow-up visit were included in this retrospective observational study.
Period: Overall Study
Arm/Group | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Started | 66 | 75
Completed | 66 | 75
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy | Total
Number analyzed (Participants) | 66 | 75 | 141
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.9 (11.8) | 57.5 (10.7) | 56.7 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 45 | 86
  Male | 25 | 30 | 55
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 7
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 62 | 72 | 134
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 64 | 69 | 133
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 6 | 8
Time since PsA diagnosis [Mean (Standard Deviation); unit: Years] — Time since PsA diagnosis as assessed at Baseline was reported. Baseline was defined as the initiation of tofacitinib anytime in between 14 December 2017 to 31 August 2023. Population: Here ''Number Analyzed'' signifies participants evaluable for the specific baseline characteristic.
  Years
    number analyzed (Participants) | 64 | 75 | 139
    (all) | 9.1 (8.9) | 8.4 (8.9) | 8.7 (8.9)
Time since onset of psoriasis (PsO) [Mean (Standard Deviation); unit: Years] — Time since onset of psoriasis as assessed at Baseline was reported. Baseline was defined as the initiation of tofacitinib anytime in between 14 December 2017 to 31 August 2023. Population: Here ''Number Analyzed'' signifies participants evaluable for the specific baseline characteristic.
  Years
    number analyzed (Participants) | 18 | 19 | 37
    (all) | 16.7 (15.6) | 19.5 (16.6) | 18.2 (16)
Comorbidity history [Count of Participants; unit: Participants] — Number of participants with comorbidities at baseline were reported. One participant may have more than 1 comorbidity. Baseline was defined as the initiation of tofacitinib anytime in between 14 December 2017 to 31 August 2023.
  Participants
    Cardiovascular disease | 11 | 6 | 17
    Hypertension | 19 | 31 | 50
    Malignancy | 5 | 6 | 11
    Anxiety | 7 | 5 | 12
    Depression | 17 | 12 | 29
    Inflammatory bowel disease | 1 | 3 | 4
    Diabetes | 11 | 12 | 23
    Uveitis | 1 | 1 | 2
    Metabolic syndrome | 35 | 40 | 75
    Psoriatic nail dystrophy | 6 | 6 | 12
    Fibromyalgia | 12 | 12 | 24
    Non-Melanoma Skin Cancer | 4 | 1 | 5
    Osteoporosis | 2 | 1 | 3
Smoking status [Count of Participants; unit: Participants] — Number of participants according to smoking status at Baseline were reported. Baseline was defined as the initiation of tofacitinib anytime in between 14 December 2017 to 31 August 2023.
  Participants
    Never smoked | 39 | 47 | 86
    Former smoker | 21 | 16 | 37
    Current smoker | 6 | 12 | 18
Work status [Count of Participants; unit: Participants] — Number of participants according to working status at Baseline were reported. Baseline was defined as the initiation of tofacitinib anytime in between 14 December 2017 to 31 August 2023.
  Participants
    Work full time | 32 | 36 | 68
    Working part-time or not working | 34 | 39 | 73
Body mass index [Mean (Standard Deviation); unit: kilogram/ metered square (^2)] — Population: Here ''Number Analyzed'' signifies participants evaluable for the specific baseline characteristic.
  kilogram/ metered square (^2)
    number analyzed (Participants) | 64 | 74 | 138
    (all) | 31.2 (6.6) | 33.9 (10.3) | 32.6 (8.8)
Insurance type [Count of Participants; unit: Participants] — Number of participants according to type of insurance were reported.
  Participants
    Private/commercial insurance | 47 | 56 | 103
    Medicare, Medicaid, or having no insurance | 19 | 19 | 38
Prior small molecule use [Count of Participants; unit: Participants] — Number of participants according to number of use of small molecule (methotrexate, leflunomide, sulfasalazine, apremilast) for treatment prior to baseline were reported. Baseline was defined as the initiation of tofacitinib anytime in between 14 December 2017 to 31 August 2023.
  Participants
    0 | 19 | 6 | 25
    1 | 25 | 39 | 64
    2 or more | 22 | 30 | 52
Prior biologic use [Count of Participants; unit: Participants] — Number of participants according to biologic use for treatment prior to baseline were reported. Biologics is a product that is produced from living organisms or contain components of living organisms. Baseline was defined as the initiation of tofacitinib anytime in between 14 December 2017 to 31 August 2023.
  Participants
    Prior Tumor necrosis factor (TNF) use: 0 | 17 | 27 | 44
    Prior Tumor necrosis factor (TNF) use: 1 | 21 | 24 | 45
    Prior Tumor necrosis factor (TNF) use: 2 or more | 28 | 24 | 52
    Prior non-TNF use: 0 | 34 | 44 | 78
    Prior non-TNF use: 1 | 16 | 24 | 40
    Prior non-TNF use: 2 or more | 16 | 7 | 23
Prednisone use [Count of Participants; unit: Participants] — Number of participants with prednisone use as assessed at Baseline were reported. Baseline was defined as the initiation of tofacitinib anytime in between 14 December 2017 to 31 August 2023.
  Participants
    Dose less than or equal to (<=) 10 milligrams (mg) | 1 | 5 | 6
    Dose greater than (>) 10 mg | 0 | 1 | 1
    No use | 65 | 69 | 134
Age at onset of psoriatic arthritis (PsA) [Mean (Standard Deviation); unit: Years] — Population: Here ''Number Analyzed'' signifies participants evaluable for the specific baseline characteristic.
  Years
    number analyzed (Participants) | 64 | 73 | 137
    (all) | 42.1 (12.3) | 44.2 (14.2) | 43.3 (13.3)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 6 Months in Tender Joint Count (68)
Description: Tender joint count (TJC) 68 is a method of assessing joint inflammation. Number of tender joints was determined by examining 68 joints and identifying the joints that were painful under pressure or to passive motion. The joints examined included the temporomandibular (n = 2), sternoclavicular (n = 2), acromioclavicular (n = 2), shoulder (n = 2), elbow (n = 2), wrist (n = 2), metacarpophalageal (n = 10), interphalangeal of thumb (n = 2), distal interphalangeal (n = 8), proximal interphalangeal (n =8), hip (n = 2), knee (n = 2), ankle mortise (n = 2), ankle tarsus (n = 2), metatarsophalangeal (n = 10), interphalangeal of great toe (n = 2), and proximal/distal interphalangeal of the toes (n = 8). Change from baseline in TJC at 6 months after tofacitinib treatment initiation was reported in this outcome measure. Baseline was defined as the date of tofacitinib treatment initiation anytime in between 14 December 2017 to 31 August 2023.
Time Frame: Baseline, 6 months after tofacitinib initiation (anytime in between 3 to 9 months); data collected and evaluated for over 23.5 months in this retrospective observational study
Population: Analysis population included all eligible participants whose data were included and observed in this study. Here, ''Number of Participants Analyzed'' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Tender joints
Groups:
- All Participants: All participants with a diagnosis of PsA/SpA who received tofacitinib on or after 14 December 2017 and had a 6-month follow-up visit were included in this retrospective observational study.
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 133 | 61 | 72
Tender joints | -2.5 (9.6) | -3.2 (10.6) | -2.0 (8.8)

2. Primary Outcome: Change From Baseline to 6 Months in Swollen Joint Count (66)
Description: Joint swelling was defined as soft tissue swelling that was detectable along the joint margins. Swollen Joint Count (SJC) was determined by examination of 66 joints and identifying when swelling was present. The joints examined included the temporomandibular (n = 2), sternoclavicular (n = 2), acromioclavicular (n = 2), shoulder (n = 2), elbow (n = 2), wrist (n = 2), metacarpophalangeal (n = 10), interphalangeal of thumb (n = 2), distal interphalangeal (n = 8), proximal interphalangeal (n = 8), knee (n = 2), ankle mortise (n = 2), ankle tarsus (n = 2), metatarsophalangeal (n = 10), interphalangeal of great toe (n = 2), and proximal/distal interphalangeal of the toes (n = 8). Change from baseline in SJC at 6 months after tofacitinib treatment initiation was reported in this outcome measure. Baseline was defined as the date of tofacitinib treatment initiation anytime in between 14 December 2017 to 31 August 2023.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Swollen joints
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 133 | 61 | 72
Swollen joints | -1.6 (4.7) | -2.2 (5.4) | -1.1 (4.0)

3. Primary Outcome: Percentage of Participants Achieving Minimal Disease Activity at 6 Month Follow-up Visit
Description: Psoriatic arthritis participant was defined as having minimal disease activity (MDA) when participant met at least 5 of following criteria: 1) tender joint count less than or equal to (<=) 1; 2) swollen joint count <= 1; 3) body surface area (BSA) <=3%; 4) patient pain VAS on 100 mm scale <= 15; where 0= 'no pain' and 100= 'pain as severe as can be imagined', higher scores indicated greater severity; 5) patient's global activity VAS on a 100 mm scale <= 20, where 0= 'lowest level of disease activity' and 100= 'highest level of disease activity', higher scores indicated greater level of disease activity; Health Assessment Questionnaire-Disability Index (HAQ-DI) score <=0.5, scale ranged from 0-3, where 0= 'normal or no difficulty' and 3= 'inability to perform', higher scores indicated more difficulty to perform; 6) tender entheseal point <= 1 using Leed's index ranged from 0-6; where 0= 'non tender' and 6= '6 tender tendon insertions', higher scores indicated more tendon insertions.
Time Frame: 6 month follow-up visit (anytime in between 3 to 9 months after tofacitinib initiation); data collected and evaluated over 23.5 months in this retrospective observational study
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 141 | 66 | 75
Percentage of participants | 17.8 [11.4 to 25.9] | 15.0 [7.5 to 27.1] | 20.7 [11.6 to 33.7]

4. Primary Outcome: Percentage of Participants With Percent Body Surface Area Score of 0% at 6 Month Follow-up Visit
Description: Four body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's full palmer hand) fitting in affected area of body region was counted. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint = 10 percent (%) for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Percent BSA for a body region = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual: arithmetic mean of % BSA of all 4 body regions, ranged from 0 to 100%. Higher % BSA = greater severity of psoriasis. Percentage of participants with % BSA score of 0% at 6-month follow-up visit were reported in this outcome measure.
Time Frame: as for outcome 3
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 141 | 66 | 75
Percentage of participants | 24.7 [16.2 to 35.0] | 27.1 [15.7 to 42.1] | 22.0 [11.1 to 38.0]

5. Primary Outcome: Percentage of Participants With Psoriatic Arthritis Disease Activity Score (PASDAS) Less Than (<) 3.2 at 6 Month Follow-up Visit
Description: PASDAS: patient global psoriatic arthritis assessment (PAA),physician global PAA, each scored on 100mm VAS,0=no disease activity(DA), 100=maximum DA, higher scores=greater DA;TJC(0-68);SJC(0-66);Leed's Enthesitis Index score ranging from 0-6;where 0=non tender,6=6 tender tendon insertions,higher scores=more tender insertions; tender dactylitic digit score ranging from 0-3 where 0=no tenderness,3=participant withdrew digit, higher scores=more tenderness; physical component summary(PCS) of short form 12(SF-12) score ranging from 0-100;where 0-20=severe physical health(PH)limitations,21-40=significant PH issues,41-60=moderate physical health,61-80=good PH,81-100=excellent PH. PASDAS total score were transformed & ranged from 0-10 where score 1.9 or less=remission,1.9-3.2=low disease activity(LDA),3.2-5.4=moderate DA,5.4 and higher=high DA, with higher scores indicating more severe disease. Percentage of participants with PASDAS score <3.2 (LDA) at 6-month follow-up visit were reported.
Time Frame: as for outcome 3
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 141 | 66 | 75
Percentage of participants | 21.8 [13.7 to 32.0] | 21.1 [10.1 to 37.8] | 22.5 [12.3 to 37.0]

6. Primary Outcome: Percentage of Participants With Resolution of Enthesitis
Description: Enthesis:site where joint capsules,ligaments,tendons attach to bone.Enthesitis is inflammation of entheses.This inflammation lead to severe pain,discomfort.Resolution of enthesitis determined by Spondyloarthritis Research Consortium of Canada(SPARCC)Enthesitis Index evaluates presence,severity of enthesitis at specific sites on body & includes:medial epicondyle,lateral epicondyle,supraspinatus insertion into greater tuberosity of humerus,greater trochanter,quadriceps insertion into superior border of patella,patellar ligament insertion into interior pole of patella/tibial tubercle,achilles tendon insertion into calcaneum,plantar fascia insertion into calcaneum.Each site is scored based on tenderness,ranged from 0-16.Higher scores=more severe enthesitis.Enthesitis was considered as resolved in those participants who had SPARCC >0 at 6 month follow-up visit(anytime in between 3-9 months after tofacitinib initiation).Percentage of participants with resolution of enthesitis were reported.
Time Frame: as for outcome 3
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 141 | 66 | 75
Percentage of participants | 35.2 [22.7 to 49.4] | 33.3 [16.4 to 55.3] | 36.7 [20.5 to 56.1]

7. Primary Outcome: Percentage of Participants With Resolution of Dactylitis
Description: Dactylitis is severe inflammation of the finger or toe tendons and joints, making them look like sausages. Resolution of dactylitis can be achieved by usage of NSAIDs, local steroid injections, biologic drugs and DMARDs. Resolution in dactylitis was considered when the following criteria were met: reduction in swelling: the affected digits showed a significant decrease in swelling; pain relief: there was a notable reduction or complete absence of pain in the affected area; improved functionality: the digits regained normal function and movement; absence of tenderness: the affected area no longer exhibited tenderness upon examination. Percentage of participants with resolution of dactylitis were reported in this outcome measure.
Time Frame: as for outcome 3
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 141 | 66 | 75
Percentage of participants | 27.8 [9.69 to 53.5] | 28.6 [5.1 to 69.7] | 27.3 [7.3 to 60.7]

8. Primary Outcome: Percentage of Participants Achieving Score of "Clear" or "Almost Clear" According to Investigator Global Assessment (IGA) of Psoriasis (PsO)
Description: The Investigator's Global Assessment (IGA) is a tool used to assess the severity of psoriasis. It is a scale that typically ranges from 0 to 4, where 0 indicates clear skin (no signs of psoriasis), 1 indicates almost clear (minimal signs of psoriasis), 2 indicates mild psoriasis, 3 indicates moderate psoriasis and 4 indicates severe psoriasis, higher scores indicated greater severity of psoriasis and provides a subjective evaluation of the overall severity of psoriasis based on clinical signs such as erythema, induration, and scaling. Percentage of participants with score of "Clear" (score 0) or "Almost Clear" (score 1) according to IGA of PsO were reported in this outcome measure.
Time Frame: as for outcome 3
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 141 | 66 | 75
Percentage of participants | 27.8 [16.5 to 41.6] | 28.6 [14.0 to 48.9] | 26.9 [12.4 to 48.1]

9. Primary Outcome: Change From Baseline at 6 Months Follow-up Visit in Disease Activity in Psoriatic Arthritis (DAPSA)
Description: DAPSA assessed the joint domain of PsA and was derived from the sum of the following components: tender joint count (0-68), swollen joint count (0-66), CRP level (milligram per deciliter [mg/dL]), participant assessment of pain (0 to 10 cm VAS, 0= no pain, 10= worst possible pain, higher scores indicated more pain), and participant's global assessment of disease activity on arthritis (0 to 10 cm VAS, 0= excellent and 10= poor, higher scores indicated more disease activity). DAPSA score ranges from 0 to more than (>) 28. Where 0-4 indicates remission, 5-14 indicates low disease activity, 15-28 indicates moderate disease activity and >28 indicates high disease activity. A higher DAPSA score indicated more active disease activity.
Time Frame: Baseline, 6 months follow-up visit after tofacitinib initiation (anytime in between 3 to 9 months); data collected and evaluated for over 23.5 months in this retrospective observational study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 69 | 27 | 42
Units on a scale | -7.2 (15.6) | -10.7 (19.3) | -4.9 (12.4)

10. Primary Outcome: Change From Baseline at 6 Months Follow-up Visit in Psoriatic Arthritis Disease Activity (PASDAS) Score
Description: PASDAS is composite PsA disease activity score that included: patient global psoriatic arthritis assessment, physician global psoriatic arthritis assessment, each scored on 100 mm VAS scale where 0= "no disease activity", 100= "maximum disease activity", higher scores indicated greater disease activity; TJC (0-68); SJC (0-66); Leed's Enthesitis Index score ranging from 0-6; where 0=non tender, 6=6 tender tendon insertions, higher scores indicated more tender insertions; tender dactylitic digit score ranging from 0-3 where 0=no tenderness, 3=participant withdrew digit, higher scores indicated more tenderness; PCS of SF-12 score ranging from 0-100; where 0-20=severe physical health limitations, 21-40=significant physical health issues, 41-60=moderate physical health, 61-80=good physical health and 81-100=excellent physical health. PASDAS total score were transformed and ranged from 0 to 10, with higher scores indicating more severe disease.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 68 | 27 | 41
Units on a scale | -1.1 (1.5) | -1.3 (1.5) | -1.0 (1.6)

11. Primary Outcome: Change From Baseline at 6 Month Follow-up Visit in Patient's Global Assessment of Pain Score (VAS)
Description: Participants self-reported assessment of the severity of their arthritis pain using a 100 mm VAS by placing a mark on the scale between 0 (no pain) and 100 (most severe pain), which corresponded to the magnitude of their pain, where higher scores indicated greater severity of pain.
Time Frame: as for outcome 9
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 141 | 66 | 75
Units on a scale | -8.9 (27.2) | -13.7 (30.0) | -4.7 (23.8)

12. Primary Outcome: Change From Baseline at 6 Month Follow-up Visit in Patient's Global Assessment of Fatigue Score (VAS)
Description: Participants self-reported assessment of the severity of their arthritis fatigue using a 100 mm VAS by placing a mark on the scale between 0 (no fatigue) and 100 (most severe fatigue), which corresponded to the magnitude of their fatigue, where higher scores indicated greater severity of fatigue.
Time Frame: as for outcome 9
Population: Analysis population included all eligible participants whose data were included and observed in this study.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 141 | 66 | 75
Units on a scale | -5.9 (24.8) | -10.8 (25.6) | -1.6 (23.5)

13. Primary Outcome: Change From Baseline at 6 Month Follow-up Visit in Investigator Global Assessment (IGA) of PsO
Description: The IGA is a tool used to assess the severity of psoriasis. It is a scale that typically ranges from 0 (clear) to 4 (severe) higher scores indicated greater severity of psoriasis and provides a subjective evaluation of the overall severity of psoriasis based on clinical signs such as erythema, induration, and scaling.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 135 | 63 | 72
Units on a scale | -0.3 (1.1) | -0.3 (1.1) | -0.2 (1.1)

14. Primary Outcome: Change From Baseline at 6 Month Follow-up Visit in Percentage Body Surface Area (BSA)
Description: Four body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's full palmer hand) fitting in affected area of a body region was counted. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint = 10% for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Percent BSA for a body region = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual: arithmetic mean of % BSA of all 4 body regions, ranged from 0 to 100%. Higher % BSA = greater severity of psoriasis.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage BSA
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 135 | 63 | 72
Percentage BSA | -0.7 (8.6) | -1.7 (8.7) | 0.2 (8.6)

15. Primary Outcome: Change From Baseline at 6 Month Follow-up Visit in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score
Description: HAQ-DI assesses the degree of difficulty a participant has experienced during the past week in 8 domains of daily living activities: dressing or grooming; arising; eating; walking; reach; grip; hygiene; and other activities. There were total of 30 items distributed in these 8 domains. Each item was scored on a 4-point scale from 0 to 3: 0= no difficulty; 1= some difficulty; 2= much difficulty; 3= unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0 (least difficulty) and 3 (extreme difficulty), where higher scores indicate more difficulty while performing daily living activities.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 139 | 64 | 75
Units on a scale | -0.1 (0.5) | -0.1 (0.4) | 0.0 (0.5)

16. Primary Outcome: Change From Baseline at 6 Month Follow-up Visit in Percentage Work Time Missed
Description: The Work Productivity and Activity Impairment (WPAI) assessed work productivity and impairment. It is a 6-item questionnaire used to assess degree to which psoriasis affected work productivity and regular activities over the past 7 days. Questions were as follows: question 1=currently employed; question 2=hours missed due to health problems; question 3=hours missed due to other reasons; question 4=hours actually worked; question 5=degree problem affected productivity while working (VAS 0-100 scale, with higher numbers indicating less productivity); question 6=degree problem affected regular activities (VAS 0-100 scale, with higher numbers indicating greater impairment of regular activities). Percent work time missed due to health problem was calculated as: question 2/ (question 2+question 4) and score ranged from 0-100% where higher numbers indicate greater impairment and less productivity. Change from baseline in percentage work time missed at 6 month follow-up visit was reported.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage work time missed
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 51 | 26 | 25
Percentage work time missed | -1.9 (15.9) | -6.1 (17.3) | 2.5 (13.1)

17. Primary Outcome: Change From Baseline at 6 Month Follow-up Visit in Percentage Impairment While Working
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which psoriasis affected work productivity and regular activities over the past 7 days. The questions are as follows: question 1 = currently employed; question 2 = hours missed due to health problems; question 3 = hours missed due to other reasons; question 4 = hours actually worked; question 5 = degree health affected productivity while working (0-10 scale, with higher numbers indicating less productivity); question 6 = degree health affected regular activities (0-10 scale, with higher numbers indicating greater impairment of regular activities). Percent impairment while working due to problem was calculated as: question 5/10 and score ranged from 0-100% where higher numbers indicate greater impairment and less productivity. Change from baseline in percentage impairment while working at 6 month follow-up visit was reported.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage impairment
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 58 | 29 | 29
Percentage impairment | -6.3 (21.7) | -12.7 (23.3) | 0.1 (18.3)

18. Primary Outcome: Change From Baseline at 6 Month Follow-up Visit in Percentage Overall Work Impairment
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which psoriasis affected work productivity and regular activities over the past 7 days. The questions are as follows: question 1 = currently employed; question 2 = hours missed due to health problems; question 3 = hours missed due to other reasons; question 4 = hours actually worked; question 5 = degree health affected productivity while working (0-10 scale, with higher numbers indicating less productivity); question 6 = degree health affected regular activities (0-10 scale, with higher numbers indicating greater impairment of regular activities). Percent overall work impairment due to problem was calculated as: question 2/ (question 2+question 4) + [(1- question 2/ (question 2+question 4) * (Q5/10)] and score ranged from 0-100% where higher numbers indicate greater impairment. Change from baseline in percentage overall work impairment at 6 month follow-up visit was reported.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage work impairment
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 51 | 26 | 25
Percentage work impairment | -6.0 (22.9) | -13.0 (20.7) | 1.4 (23.1)

19. Primary Outcome: Change From Baseline at 6 Month Follow-up Visit in Percentage Activity Impairment
Description: The WPAI assesses work productivity and impairment. It is a 6-item questionnaire used to assess the degree to which psoriasis affected work productivity and regular activities over the past 7 days. The questions are as follows: question 1 = currently employed; question 2 = hours missed due to health problems; question 3 = hours missed due to other reasons; question 4 = hours actually worked; question 5 = degree health affected productivity while working (0-10 scale, with higher numbers indicating less productivity); question 6 = degree health affected regular activities (0-10 scale, with higher numbers indicating greater impairment of regular activities). Percent activity impairment due to problem was calculated as: question 6/10 and score ranged from 0-100% where higher numbers indicate greater impairment. Change from baseline in percentage activity impairment at 6 month follow-up visit was reported.
Time Frame: as for outcome 9
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage activity impairment
Arm/Group | All Participants | Tofacitinib Monotherapy | Tofacitinib + OSM Combination Therapy
Number analyzed (Participants) | 60 | 29 | 31
Percentage activity impairment | -12.1 (25.8) | -21.8 (28.9) | -2.9 (18.7)

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not collected during the study.
Description: In this observational retrospective study of deidentified database individual identifying information was not available. Minimum criteria for reporting an adverse event could not be met, hence serious adverse events (SAEs) and other adverse events (AEs) were not collected and reported.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/14/NCT05195814/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/14/NCT05195814/SAP_001.pdf